CLINICAL TRIAL: NCT03535701
Title: Ketogenic Diet and Chemotherapy to Affect Recurrence of Breast Cancer (The KETO-CARE Study)
Brief Title: Ketogenic Diet and Chemotherapy in Affecting Recurrence in Patients With Stage IV Breast Cancer
Acronym: KETO-CARE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Jeff Volek, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-16289; NCI-2017-01168 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-05-09; First posted 2018-05-24 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: interventions — Diet Therapy; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (standard of care) (Active Comparator): Patients receive standard of care therapy with paclitaxel.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (standard of care, ketogenic diet) (Experimental): Patients receive standard of care with paclitaxel. Patients undergo a controlled feeding period ketogenic diet comprising of meals prepared in the research kitchen for 3 months. Beginning 2 weeks prior to completion of the controlled feeding period, patients also undergo free living ketogenic diet program for 3 months comprising of group format, individual sessions, and online digital content to educate patients to implement a ketogenic eating pattern into their lifestyle.
  Interventions: Dietary Supplement: Dietary Intervention; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Dietary Supplement: Dietary Intervention — Undergo ketogenic diet
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Arm II (standard of care, ketogenic diet)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given standard of care therapy with paclitaxel
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies how well a ketogenic diet and chemotherapy work in affecting the return of cancer in patients with stage IV breast cancer. Ketogenic diet may be more effective than standard nutrition and may affect quality of life, inflammation, and tumor-related changes. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ketogenic diet and chemotherapy may be better in patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of implementing a diet that induces nutritional ketosis in women who are initiating palliative chemotherapy to treat advanced stage breast cancer (BC).

II. To determine the effects of a ketogenic diet on tumor progression. III. To determine the effects of nutritional ketosis on biologic and behavioral health markers.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I: Patients receive standard of care therapy with paclitaxel.

ARM II: Patients receive standard of care with paclitaxel. Patients undergo a controlled feeding period ketogenic diet comprising of meals prepared in the research kitchen for 3 months. Beginning 2 weeks prior to completion of the controlled feeding period, patients also undergo free living ketogenic diet program for 3 months comprising of group format, individual sessions, and online digital content to educate patients to implement a ketogenic eating pattern into their lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) >= 22 kg/m^2
* Confirmed diagnosis of metastatic or stage IV BC
* Fludeoxyglucose F-18 (FDG)-positron emission tomography (PET) avid tumors
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (0=participant has either normal activity, 1= participant has some symptoms but is nearly full ambulatory)
* Life expectancy > 6 months
* Able and willing to follow prescribed diet intervention

Exclusion Criteria:

* Prior chemotherapy for metastatic breast cancer (MBC) (prior adjuvant chemotherapy permitted as long as > 12 months [mo])
* BMI < 25 kg/m^2
* Weight change > 5% within 3 months of enrollment
* Type 1 diabetes
* History of diabetes with retinopathy requiring treatment
* Current use of insulin or sulfonylureads for glycemic control, or history of ketoacidosis
* Intestinal obstruction
* Bilirubin > 2
* Albumin < 3.5
* Glomerular filtration rate (GFR) < 55 mL/min
* Creatinine > 2.0
* Urinary albumin > 1 g/day
* Congestive heart failure
* Pregnant or nursing women
* Unable to provide informed consent
* Uncontrolled concurrent medical conditions that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Adherence and compliance to the ketogenic diet | Up to 26 weeks
  Summaries from diet assessments and ketone logs will be plotted over time to assess adherence and compliance to the ketogenic diet.
Changes in psychosocial measures | Baseline up to 26 weeks
  Summary measures such as Cohens d will be used. Linear and nonlinear mixed models will be used as appropriate to model changes in tumor markers, comorbidity risk factors, and other measures over time, with emphasis will be on estimating effect sizes (such as slopes of change). Post hoc tests will be used to examine pairwise comparisons when significant main or interaction effects are observed. The alpha level for significance will be set at p =< 0.05.
Changes in physiologic outcomes | Baseline up to 26 weeks
  Summary measures such as Cohens d will be used. Linear and nonlinear mixed models will be used as appropriate to model changes in tumor markers, comorbidity risk factors, and other measures over time, with emphasis will be on estimating effect sizes (such as slopes of change). Post hoc tests will be used to examine pairwise comparisons when significant main or interaction effects are observed. The alpha level for significance will be set at p =< 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Volek, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu